CLINICAL TRIAL: NCT06023368
Title: Reducing Port Access Pain and Clinic Wait Time: An Evaluation of EMLA Cream Versus nüm™ Vapocoolant Spray
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Administrative burden
Sponsor: Marianne Hutti (Other)
Collaborators: Bimeco Group (Unknown)
Responsible Party: Sponsor-Investigator, Marianne Hutti, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 84569
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Pediatric Cancer
Keywords: Port access pain; pediatric; oncology
MeSH Terms: conditions — Neoplasms | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sterile Vapocoolant Spray (Experimental): Num vapocoolant spray will be administered as a single use canister around the port
  Interventions: Drug: Num Vapocoolant Spray
- EMLA Cream (Active Comparator): Numbing (EMLA) cream will be applied around the port.
  Interventions: Drug: EMLA Cream

INTERVENTIONS:
Drug: Num Vapocoolant Spray — Spray applied around port prior to access
  Other Names: Vapocoolant Spray
  Arms: Sterile Vapocoolant Spray
Drug: EMLA Cream — cream applied around the port prior to access
  Other Names: numbing cream
  Arms: EMLA Cream

SUMMARY:
The goal of this clinical trial is to compare a sterile vapocoolant spray to EMLA cream in children with access ports.

Participants will receive either the spray or cream prior to port access and rate pain on a scale.

Researchers will compare spray vs cream to see if the spray is as effective as the cream in reducing pain associated with port puncture.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Present appointment is for drawing blood, receiving intravenous antibiotics, blood products, or chemotherapy
* EMLA cream has (standard of care) or has not (vapocoolant) been applied to the port site prior to the appointment
* Previous allergic reaction or skin irritation due to EMLA
* Quick access to the child's port is needed for drawing blood, or giving treatments, blood products, or drugs such as chemotherapy

Exclusion Criteria:

* Child has a legal guardian or non-parent family member as the only adult with them for the visit.
* Children less than 4 years of age
* Children with altered mental status
* History of traumatic brain injury, developmental delay or autism
* Child is nonverbal
* Present appointment is for drawing blood, receiving intravenous antibiotics, blood products, or chemotherapy, and child and parents prefer to wait for EMLA cream to take effect.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-23 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Port Access Pain | Within 5 minutes of port access
  Pain will be measured by The Faces Pain Scale - Revised (FPS-R). FPS-R is a self-report measure of pain intensity developed for children. It was adapted from the Faces Pain Scale to make it possible to score the sensation of pain on the widely accepted 0-to-10 metric. Higher scores mean increased pain.
Clinic Wait Time | Day of visit, up to 8 hours
  Wait time will be measured in minutes from check in to check out
Duration of Visit | Day of visit, up to 8 hours
  Total length of overall appointment time measured in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Hutti, PhD, APRN, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky DanceBlue Pediatric Hematology/oncology clinic, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No